CLINICAL TRIAL: NCT00579800
Title: Newer Breast MRI Sequences for the Evaluation of Breast Cancer -FIESTA, Vibrant-DE and IDEAL: Feasibility Evaluation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 07-091; NCT00514319 (obsolete NCT alias)
Record Dates: First submitted 2007-12-20; First posted 2007-12-24 (Estimated); Last update posted 2016-05-10 (Estimated); Status verified 2016-05

CONDITIONS: Breast Cancer
Keywords: Vibrant-DE; IDEAL; MRI; Breast; 07-091
MeSH Terms: conditions — Breast Neoplasms

ARMS (1):
- women undergoing routine breast MRI (Experimental): Conventional images will be taken using the standard sequences consisting of T2-weighted imaging and T1-weighted imaging before and after contrast; these will be used for the diagnostic examination. FIESTA will be performed on 50 patients, while Vibrant-DE and IDEAL will be performed on the other 50 patients.
  Interventions: Procedure: new software sequences, FIESTA and Vibrant-DE and IDEAL

INTERVENTIONS:
Procedure: new software sequences, FIESTA and Vibrant-DE and IDEAL — Conventional images will be taken using the standard sequences consisting of T2-weighted imaging and T1-weighted imaging before and after contrast; these will be used for the diagnostic examination. FIESTA will be performed on 50 patients, while Vibrant-DE and IDEAL will be performed on the other 50 patients.

SUMMARY:
The purpose of this study is to evaluate new computer software on breast magnetic resonance imaging (MRI). The information from this study may help doctors and scientists develop better ways to find breast cancer, and may help future patents with cancer.

ELIGIBILITY:
Inclusion Criteria:

* Female patients over the age of 21 undergoing a diagnostic Breast MRI.

Exclusion Criteria:

* Patients who would be normally excluded from undergoing an MRI examination
* Patients with a pacemaker, aneurysm clip or any other condition that would warrant avoidance of a strong magnetic field.
* Patients under the age of 21.
* Female patients who are pregnant.

Min Age: 21 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2007-07; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
To evaluate the feasibility of three new pulse sequences for breast MRI using newly developed software; FIESTA, Vibrant DE and IDEAL | conclusion of the study

SECONDARY OUTCOMES:
To quantitatively and qualitatively assess performance of the three breast pulse sequences, and compare these results with the same parameters on standard breast MRI sequences. | conclusion of the study

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Morris, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan Kettering Web Site — http://www.mskcc.org